CLINICAL TRIAL: NCT02604849
Title: Efficacy of Intestinal Decontamination in Patients Colonized by Carbapenem-resistant Klebsiella Pneumoniae and Colistin
Status: Completed | Type: Observational
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Other Study IDs: FCO-NEE-2015-01
Record Dates: First submitted 2015-11-10; First posted 2015-11-13 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Patients Colonized by Klebsiella Pneumoniae.
MeSH Terms: interventions — Neomycin; Streptomycin; Gentamicins

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Received therapy desconolizacion against Klebsiella pneumoniae
  Interventions: Drug: Neomycin; Drug: Streptomycin; Drug: Gentamicins
- Patients who do not receive the therapy

INTERVENTIONS:
Drug: Neomycin
  Groups: Received therapy desconolizacion against Klebsiella pneumoniae
Drug: Streptomycin
  Groups: Received therapy desconolizacion against Klebsiella pneumoniae
Drug: Gentamicins
  Groups: Received therapy desconolizacion against Klebsiella pneumoniae

SUMMARY:
The identification of all cases (44 patients) was carried out from the database of microbiology, University Hospital Reina Sofía and the University Hospital of Jerez. For the identification of controls, in case of neutropenic patients, all colonized patients that were included during the study period did not receive any decolonitation treatment; in case of non-neutropenic patients it was studied a paired control by the presence of risk factors that indicated the beginning of decolonitation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with intestinal colonization by Klebsiella pneumoniae, defined as the presence of a positive rectal swab culture at least 7 days prior to initiation of therapy; and patients considered at risk of developing an invasive infection by Klebsiella pneumoniae:
* Surgery in two weeks
* Transplant in two weeks
* Require medical intervention or has a clinical situation that may predispose to the development of a serious infection (chemotherapy, immunosuppression or neutropenia)
* Recurrent or severe infections
* Institution admission
* Fragile patients at high risk of readmission.

Exclusion Criteria:

* The presence of an active infection for Klebsiella Pneumoniae.
* Concomitant use of systemic antibiotics in the 14 days before the start of decolonization therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample consists of all patients who received therapy desconolizacion against Klebsiella Pneumoniae versus those not receiving such therapy.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2012-07; Primary Completion 2015-07 (Actual); Study Completion 2015-11

PRIMARY OUTCOMES:
Mortality for any cause during a six-months period after oral therapy gut decontamination. | 6 months

REFERENCES:
- [Derived] Machuca I, Gutierrez-Gutierrez B, Perez Cortes S, Gracia-Ahufinger I, Serrano J, Madrigal MD, Barcala J, Rodriguez-Lopez F, Rodriguez-Bano J, Torre-Cisneros J. Oral decontamination with aminoglycosides is associated with lower risk of mortality and infections in high-risk patients colonized with colistin-resistant, KPC-producing Klebsiella pneumoniae. J Antimicrob Chemother. 2016 Nov;71(11):3242-3249. doi: 10.1093/jac/dkw272. Epub 2016 Jul 26. PMID 27494911